CLINICAL TRIAL: NCT02208349
Title: King Video Laryngoscope Versus Direct Laryngoscopy for Prehospital Intubation: A Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis suggested additional enrollment would not change outcomes
Sponsor: Saint Vincent Hospital, Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LECOM Research Grant 2013
Record Dates: First submitted 2014-03-18; First posted 2014-08-05 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Respiratory Failure
Keywords: intubation, laryngoscopy, prehospital, emergency medical services
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Video Laryngoscopy (Experimental): We will outfit ½ of the ambulance crews with the King Video Laryngoscope (KVL) for 6 months while the other ½ of the ambulances will use traditional direct laryngoscopy (DL). After 6 months, the groups will switch devices. We will randomly assign those ambulances that first use the KVL. After one year (12 months) we will compare the outcomes between the two methods.
  Interventions: Device: King Video Laryngoscope
- Direct Laryngoscopy (Active Comparator): We will outfit ½ of the ambulance crews with the King Video Laryngoscope (KVL) for 6 months while the other ½ of the ambulances will use traditional direct laryngoscopy (DL). After 6 months, the groups will switch devices. We will randomly assign those ambulances that first use the KVL. After one year (12 months) we will compare the outcomes between the two methods.
  Interventions: Device: traditional direct laryngoscopy (DL)

INTERVENTIONS:
Device: King Video Laryngoscope — We will outfit ½ of the ambulance crews with the King Video Laryngoscope (KVL) for 6 months while the other ½ of the ambulances will use traditional direct laryngoscopy (DL). After 6 months, the groups will switch devices. We will randomly assign those ambulances that first use the KVL. After one year (12 months) we will compare the outcomes between the two methods.
  Arms: Video Laryngoscopy
Device: traditional direct laryngoscopy (DL)
  Arms: Direct Laryngoscopy

SUMMARY:
The goal of this study is to compare the first pass success rate of intubation between video assisted intubation and traditional direct visualization intubation in the field by Emergency Medical Service (EMS) professionals

DETAILED DESCRIPTION:
We will equip several local advanced life support ambulances with a low cost video laryngoscope for a total of 12 months. We will outfit ½ of the ambulance crews with the King Video Laryngoscope (KVL) for 6 months while the other ½ of the ambulances will use traditional direct laryngoscopy (DL). After 6 months, the groups will switch devices. We will randomly assign those ambulances that first use the KVL. After one year (12 months) we will compare the outcomes between the two methods including first pass intubation success, total success rate for intubation, and complications (need for surgical airway, rescue device, need to revert from KVL to DL, etc.). Please see the attached protocol page for additional details.

ELIGIBILITY:
Inclusion Criteria:

* all patients >= age 18 year of age undergoing ETI in the prehospital setting

Exclusion Criteria:

* age < 18 years of age

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Vincent Hospital, Erie, Pennsylvania, United States

REFERENCES:
- [Background] Pepe PE, Copass MK, Joyce TH. Prehospital endotracheal intubation: rationale for training emergency medical personnel. Ann Emerg Med. 1985 Nov;14(11):1085-92. doi: 10.1016/s0196-0644(85)80927-6. PMID 3931512
- [Background] Wang HE, Mann NC, Mears G, Jacobson K, Yealy DM. Out-of-hospital airway management in the United States. Resuscitation. 2011 Apr;82(4):378-85. doi: 10.1016/j.resuscitation.2010.12.014. Epub 2011 Feb 1. PMID 21288624
- [Background] Mort TC. Emergency tracheal intubation: complications associated with repeated laryngoscopic attempts. Anesth Analg. 2004 Aug;99(2):607-13, table of contents. doi: 10.1213/01.ANE.0000122825.04923.15. PMID 15271750
- [Background] Katz SH, Falk JL. Misplaced endotracheal tubes by paramedics in an urban emergency medical services system. Ann Emerg Med. 2001 Jan;37(1):32-7. doi: 10.1067/mem.2001.112098. PMID 11145768
- [Background] Jones JH, Murphy MP, Dickson RL, Somerville GG, Brizendine EJ. Emergency physician-verified out-of-hospital intubation: miss rates by paramedics. Acad Emerg Med. 2004 Jun;11(6):707-9. doi: 10.1197/j.aem.2003.12.026. PMID 15175215
- [Background] Hubble MW, Brown L, Wilfong DA, Hertelendy A, Benner RW, Richards ME. A meta-analysis of prehospital airway control techniques part I: orotracheal and nasotracheal intubation success rates. Prehosp Emerg Care. 2010 Jul-Sep;14(3):377-401. doi: 10.3109/10903121003790173. PMID 20507222
- [Background] Wang HE, Yealy DM. How many attempts are required to accomplish out-of-hospital endotracheal intubation? Acad Emerg Med. 2006 Apr;13(4):372-7. doi: 10.1197/j.aem.2005.11.001. Epub 2006 Mar 10. PMID 16531595
- [Background] Lossius HM, Roislien J, Lockey DJ. Patient safety in pre-hospital emergency tracheal intubation: a comprehensive meta-analysis of the intubation success rates of EMS providers. Crit Care. 2012 Feb 11;16(1):R24. doi: 10.1186/cc11189. PMID 22325973
- [Background] Warner KJ, Carlbom D, Cooke CR, Bulger EM, Copass MK, Sharar SR. Paramedic training for proficient prehospital endotracheal intubation. Prehosp Emerg Care. 2010 Jan-Mar;14(1):103-8. doi: 10.3109/10903120903144858. PMID 19947874
- [Background] Carlson JN, Quintero J, Guyette FX, Callaway CW, Menegazzi JJ. Variables associated with successful intubation attempts using video laryngoscopy: a preliminary report in a helicopter emergency medical service. Prehosp Emerg Care. 2012 Apr-Jun;16(2):293-8. doi: 10.3109/10903127.2011.640764. Epub 2011 Dec 22. PMID 22191806
- [Background] Guyette FX, Farrell K, Carlson JN, Callaway CW, Phrampus P. Comparison of video laryngoscopy and direct laryngoscopy in a critical care transport service. Prehosp Emerg Care. 2013 Apr-Jun;17(2):149-54. doi: 10.3109/10903127.2012.729128. Epub 2012 Dec 11. PMID 23231426
- [Background] Sakles JC, Mosier J, Chiu S, Cosentino M, Kalin L. A comparison of the C-MAC video laryngoscope to the Macintosh direct laryngoscope for intubation in the emergency department. Ann Emerg Med. 2012 Dec;60(6):739-48. doi: 10.1016/j.annemergmed.2012.03.031. Epub 2012 May 5. PMID 22560464
- [Background] Mosier JM, Stolz U, Chiu S, Sakles JC. Difficult airway management in the emergency department: GlideScope videolaryngoscopy compared to direct laryngoscopy. J Emerg Med. 2012 Jun;42(6):629-34. doi: 10.1016/j.jemermed.2011.06.007. Epub 2011 Sep 10. PMID 21911279
- [Background] Wayne MA, McDonnell M. Comparison of traditional versus video laryngoscopy in out-of-hospital tracheal intubation. Prehosp Emerg Care. 2010 Apr-Jun;14(2):278-82. doi: 10.3109/10903120903537189. PMID 20199237
- [Background] Akihisa Y, Maruyama K, Koyama Y, Yamada R, Ogura A, Andoh T. Comparison of intubation performance between the King Vision and Macintosh laryngoscopes in novice personnel: a randomized, crossover manikin study. J Anesth. 2014 Feb;28(1):51-7. doi: 10.1007/s00540-013-1666-9. Epub 2013 Jun 30. PMID 23812581

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 83 were enrolled and 82 met inclusion criteria.
Units Other Than Participants: Ambulance
Groups:
- Video Laryngoscopy First Then Direct Laryngoscopy: We will outfit ½ of the ambulance crews with the King Video Laryngoscope (KVL) for 6 months while the other ½ of the ambulances will use traditional direct laryngoscopy (DL). After 6 months, the groups will switch devices. We will randomly assign those ambulances that first use the KVL. After one year (12 months) we will compare the outcomes between the two methods.
  King Video Laryngoscope: We will outfit ½ of the ambulance crews with the King Video Laryngoscope (KVL) for 6 months while the other ½ of the ambulances will use traditional direct laryngoscopy (DL). After 6 months, the groups will switch devices. We will randomly assign those ambulances that first use the KVL. After one year (12 months) we will compare the outcomes between the two methods.
- Direct Laryngoscopy First Then Video Laryngoscopy: We will outfit ½ of the ambulance crews with the King Video Laryngoscope (KVL) for 6 months while the other ½ of the ambulances will use traditional direct laryngoscopy (DL). After 6 months, the groups will switch devices. We will randomly assign those ambulances that first use the KVL. After one year (12 months) we will compare the outcomes between the two methods.
  traditional direct laryngoscopy (DL)
Period: Initial 6 Months
Arm/Group | Video Laryngoscopy First Then Direct Laryngoscopy | Direct Laryngoscopy First Then Video Laryngoscopy
Started | 16; 3 Ambulance | 9; 3 Ambulance
Completed | 16; 3 Ambulance | 9; 3 Ambulance
Not Completed | 0; 0 Ambulance | 0; 0 Ambulance
Period: Second 6 Months
Arm/Group | Video Laryngoscopy First Then Direct Laryngoscopy | Direct Laryngoscopy First Then Video Laryngoscopy
Started | 11; 3 Ambulance | 7; 3 Ambulance
Completed | 11; 3 Ambulance | 7; 3 Ambulance
Not Completed | 0; 0 Ambulance | 0; 0 Ambulance
Period: Third 6 Month
Arm/Group | Video Laryngoscopy First Then Direct Laryngoscopy | Direct Laryngoscopy First Then Video Laryngoscopy
Started | 6; 3 Ambulance | 3; 3 Ambulance
Completed | 6; 3 Ambulance | 3; 3 Ambulance
Not Completed | 0; 0 Ambulance | 0; 0 Ambulance
Period: Fourth 6 Month
Arm/Group | Video Laryngoscopy First Then Direct Laryngoscopy | Direct Laryngoscopy First Then Video Laryngoscopy
Started | 14; 3 Ambulance | 2; 3 Ambulance
Completed | 14; 3 Ambulance | 2; 3 Ambulance
Not Completed | 0; 0 Ambulance | 0; 0 Ambulance
Period: Fifth 6 Month
Arm/Group | Video Laryngoscopy First Then Direct Laryngoscopy | Direct Laryngoscopy First Then Video Laryngoscopy
Started | 7; 3 Ambulance | 2; 3 Ambulance
Completed | 7; 3 Ambulance | 2; 3 Ambulance
Not Completed | 0; 0 Ambulance | 0; 0 Ambulance
Period: Sixth 6 Month
Arm/Group | Video Laryngoscopy First Then Direct Laryngoscopy | Direct Laryngoscopy First Then Video Laryngoscopy
Started | 3; 3 Ambulance | 2; 3 Ambulance
Completed | 3; 3 Ambulance | 2; 3 Ambulance
Not Completed | 0; 0 Ambulance | 0; 0 Ambulance

BASELINE CHARACTERISTICS:
Groups:
- Video Laryngoscopy Treatment: Patients treated by ambulance agency with video laryngoscopy.
- Direct Laryngoscopy Treatment: Patients treated by ambulance agency with direct laryngoscopy.
- Total: Total of all reporting groups
Arm/Group | Video Laryngoscopy Treatment | Direct Laryngoscopy Treatment | Total
Number analyzed (Participants) | 40 | 42 | 82
Age, Customized [Count of Participants; unit: Participants]
  Age 18-59 | 11 | 13 | 24
  Age 60 and over | 29 | 29 | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 28 | 33 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful First Intubation Attempt (First Pass Attempt)
Description: Endotracheal Intubation (ETI) attempt will be defined as tip of the laryngoscope blade passing the patient's lips. First attempt success rate will be defined as the number of successful placements occurring on the first attempt to place the endotracheal tube.
Time Frame: less than 24 hours, collected for the duration of the study (approximately 34 months)
Measure: Count of Participants; unit: Participants
Groups:
- Video Laryngoscopy: Participants who were treated by an ambulance agency randomized to received VL
- Direct Laryngoscopy: Participants who were treated by an ambulance agency randomized to receive DL
Arm/Group | Video Laryngoscopy | Direct Laryngoscopy
Number analyzed (Participants) | 40 | 42
Participants | 25 | 28

2. Secondary Outcome: Overall Success
Description: Overall success rate will be defined as the total number of successful placements divided by the total number of patients treated.
Time Frame: up to 24 hours, duration of the study (approximately 34 months)
Measure: Count of Participants; unit: Participants
Groups:
- Video Laryngoscopy: Patients treated by an ambulance agency randomized to VL
- Direct Laryngoscopy: Patients treated by an ambulance agency randomized to DL
Arm/Group | Video Laryngoscopy | Direct Laryngoscopy
Number analyzed (Participants) | 40 | 42
Participants | 29 | 34

ADVERSE EVENTS:
Arm/Group | Video Laryngoscopy | Direct Laryngoscopy
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42
Other Adverse Events (participants affected / at risk) | 0/40 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Video Laryngoscopy (N=40) | Direct Laryngoscopy (N=42)
Esophageal Intubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Recognized Esophageal Intubation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No